CLINICAL TRIAL: NCT01219335
Title: Laboratory Evaluation of De-identified, Developmentally Arrested Embryos of Embryos Diagnosed as Having an Abnormal Number of Chromosomes for Optimization of Techniques for Assisted Reproduction
Brief Title: Discarded Materials Study
Status: Recruiting | Type: Observational
Sponsor: Reproductive Medicine Associates of New Jersey (Other)
Responsible Party: Sponsor
Other Study IDs: RMA-00-02
Record Dates: First submitted 2010-10-08; First posted 2010-10-13 (Estimated); Last update posted 2025-02-07 (Actual); Status verified 2025-02

CONDITIONS: Infertility
Keywords: IVF
MeSH Terms: conditions — Infertility

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Discarded non-viable oocytes, granulosa cells, spermatozoa, developmentally arrested embryos, serum, follicular fluid, and conditioned IVF media.
Oversight: Data Monitoring Committee: No

SUMMARY:
Use of discarded embryos to advance laboratory expertise and technology in the area of human embryo development and assisted reproductive technologies

DETAILED DESCRIPTION:
1- Testing methods or freezing before implementing techniques. 2- Develop cell surgery and micromanipulation techniques. 3- Develop methods to optimize the determinations of genes and chromosomes 4- Quality-assess laboratory equipment. 5- Test proficiency of laboratory staff. 6- Analyze what effects the early development of embryos. 7- Develop new methods and media to allow for higher survival rates of embryos. 8- Develop non-invasive tests for predicting embryo quality to predict IVF success.

ELIGIBILITY:
Inclusion Criteria:

none

Exclusion Criteria:

none

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: All patients undergoing infertility treatment
Sampling Method: Non-Probability Sample
Enrollment: 10000 (Estimated)
Dates: Start 2003-04; Primary Completion 2025-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Methods for freezing -embryos | duration of the study
  To test, standardize and implement better methods for the freezing embryos prior to these techniques being used in the clinical setting

SECONDARY OUTCOMES:
Development non-invasive tests | duration of the study
  To develop non-invasive tests for predicting embryo quality as well as IVF success
Factors that control embryo development | duration of the study
  To analyze embryos to learn more about what controls their early development and function.

CONTACTS AND LOCATIONS:
Overall Officials: Thomas Molinaro, MD, MSCE, Principal Investigator — Reproductive Medicine Associates of New Jersey
Locations (1):
- Reproductive Medicine Associates of new Jersey, Basking Ridge, New Jersey, United States